CLINICAL TRIAL: NCT00760461
Title: Domperidone in Refractory Gastroparesis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Enrolled subjects were unable to receive drug from dispensing pharmacy.
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0809004202
Record Dates: First submitted 2008-09-24; First posted 2008-09-26 (Estimated); Results first posted 2017-08-18 (Actual); Last update posted 2017-08-18 (Actual); Status verified 2017-02

CONDITIONS: Gastroparesis
MeSH Terms: conditions — Gastroparesis | interventions — Domperidone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Domperidone (Other)
  Interventions: Drug: Domperidone

INTERVENTIONS:
Drug: Domperidone — 10 mg 4 times daily 20 mg 4 times daily 30 mg 4 times daily

SUMMARY:
The primary objective of this study is to prescribe oral domperidone for patients with gastroparesis who have failed or suffered adverse effects from standard medical therapy.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Age 18 and older
* Symptoms or manifestations secondary to motility disorders of the upper GI tract. These include gastroparesis, functional dyspepsia, gastroesophageal reflux disease that are refractory to standard therapy.
* Patients must have a comprehensive evaluation to eliminate other causes of their symptoms. This includes a history and physical examination. A recent (within 3 years) evaluation of the upper GI tract with either upper endoscopy or upper GI radiographic series. Baseline blood tests suggested are electrolytes, magnesium, and prolactin level.
* Patient has signed informed consent for the administration of domperidone that informs the patient of potential adverse events including:

  * Increased prolactin levels
  * Breast changes
  * Extrapyramidal side effects
  * Cardiac arrhythmias including QT prolongation (increased risk with the drugs listed in the appendix)

Exclusion Criteria:

* History of, or current, arrhythmias including ventricular tachycardia, ventricular fibrillation and Torsade des Pointes. Patients with minor forms of ectopy (PACs) are not necessarily excluded.
* Clinically significant bradycardia, sinus node dysfunction, or heart block. Prolonged QTc (QTc>450 milliseconds for males, QTc>470 milliseconds for females)
* Clinically significant electrolyte disorders. These include significant hypokalemia, hyperkalemia, hypomagnesemia, and hypermagnesemia that cannot be corrected with treatment of these electrolyte abnormalities.
* Gastrointestinal hemorrhage or obstruction.
* Presence of a prolactinoma (prolactin-releasing pituitary tumor).
* Pregnant or breast feedings female.
* Known allergy to domperidone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2008-10; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anish A Sheth, MD, Principal Investigator — Yale University
Locations (1):
- Yale Digestive Diseases 40 Temple St, Suite 1A, New Haven, Connecticut, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Domperidone
Started | 44
Completed | 0
Not Completed | 44

BASELINE CHARACTERISTICS:
Arm/Group | Domperidone
Number analyzed (Participants) | 44
Age, Categorical [Count of Participants; unit: Participants] — Age was not collected and summarized. Population: Age was not collected and summarized.
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35
  Male | 9

OUTCOME MEASURES:

1. Primary Outcome: Gastroparesis Cardinal Symptom Index
Time Frame: upon study completion
Population: Data cannot be summarized or analyzed due to the lack of data being collected on the primary outcome due to the trial being terminated.
Arm/Group | Domperidone
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Domperidone
Serious Adverse Events (participants affected / at risk) | 0/44
Other Adverse Events (participants affected / at risk) | 0/44

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes